CLINICAL TRIAL: NCT01780311
Title: Catheter Ablation Versus Antiarrhythmic Drugs for Outflow Tract Ventricular ARrhythmias
Acronym: AVATAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Other Study IDs: Arezzo008
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Ventricular Tachycardia; Ventricular Premature Complexes
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes | interventions — Anti-Arrhythmia Agents; Flecainide; Propafenone; Sotalol; Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antiarrhythmic drugs (Active Comparator): Flecainide or Propafenone or Sotalol (oral, standard dosage)
  Interventions: Drug: antiarrhythmic drugs (Flecainide or Propafenone or Sotalol)
- ABLATION (Experimental): Catheter Ablation
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Drug: antiarrhythmic drugs (Flecainide or Propafenone or Sotalol)
  Arms: Antiarrhythmic drugs
Procedure: Catheter Ablation
  Arms: ABLATION

SUMMARY:
A randomized, parallel, open study comparing catheter ablation versus antiarrhythmic drugs for outflow tract ventricular arrhythmias

ELIGIBILITY:
Inclusion Criteria:

1. presence of ventricular ectopic beats (VEB) with left-bundle-branch block morphology or right-bundle-branch block morphology and positive concordance throughout the chest leads, inferior axis and at least one of the following:

1. >2000 isolated VEB/24h
2. symptomatic monomorphic ventricular tachycardia
3. left ventricular disfunction supposed to be due to tachycardia-induced cardiomyopathy

Exclusion Criteria:

1. known structural heart disease
2. pregnancy
3. life expectancy < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 score | 6 months
  Quality of life improvement according to SF-36 score variations

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy